CLINICAL TRIAL: NCT07090850
Title: Innovative Approaches in Medical Education: The Impact of Puzzles on Learning and Motivation
Brief Title: The Impact of Puzzles on Learning and Motivation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tarsus University (Other)
Responsible Party: Principal Investigator, Nadiye BARIŞ EREN, Asst. Prof., Tarsus University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: TarsusU-NBARISEREN-005
Record Dates: First submitted 2025-07-21; First posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Education Nursing
Keywords: Nursing education; puzzle; academic achievement; motivation; randomized controlled trial

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Puzzle education group (Experimental): In the first stage, all students were explained about the research, and their consent was obtained. "Personal Information Form" was filled in by the students whose informed consents were obtained and who agreed to participate in the study under observation in the classroom environment. Then, the "Achievement Test 1" and the "IMTS" were administered to all students as a pretest. In the second stage, Roper Logan and Tierney's Life Model for Life Activities was taught interactively to all students by the same instructors for 2 hours for 1 week. The puzzle booklet previously created for this study was used in the third stage. The researchers made this booklet. In the fifth stage, "Achievement Test 2" was administered to the students in both the intervention and control groups 1 week after the training, and "IMTS" was administered as a post-test.
  Interventions: Behavioral: Puzzle education group
- Control Group (No Intervention): In the first stage, all students were explained about the research, and their consent was obtained. "Personal Information Form" was filled in by the students whose informed consents were obtained and who agreed to participate in the study under observation in the classroom environment. Then, the "Achievement Test 1" and the "IMTS" were administered to all students as a pretest. In the second stage, Roper Logan and Tierney's Life Model for Life Activities was taught interactively to all students by the same instructors for 2 hours for 1 week. In the Control Group (Branch A), routine lecturing continued without intervention in the fourth stage. In the fifth stage, "Achievement Test 2" was administered to the students in both the intervention and control groups 1 week after the training, and "IMTS" was administered as a post-test.

INTERVENTIONS:
Behavioral: Puzzle education group — It was evaluated the effect of using puzzles as a teaching technique in a nursing practice course.
  Arms: Puzzle education group

SUMMARY:
Innovative and interactive techniques are increasingly needed in nursing education to enhance students' comprehension and motivation. Puzzles are among the creative tools that may contribute to improved learning outcomes. This research offers practical implications for enhancing curriculum design and teaching practices in nursing education. This situation is aimed at increasing students' participation and motivation in the course.

Research Questions:

1. Does the use of puzzles in nursing education improve students' academic achievement?
2. Does the use of puzzles enhance students' motivation towards instructional materials?

DETAILED DESCRIPTION:
There are minimal studies on the use of puzzles in the literature. On the other hand, the importance of using puzzles as a teaching technique in education is increasing daily. This study evaluated the effect of using puzzles as a teaching technique in a nursing practice course. Despite the increasing importance of using puzzles in education, the limited research in nursing education shows the gap in this field. Especially with this technique, the student's knowledge level is expected to increase, and learning will be permanent in a critically important course in which nursing practices are taught. On the other hand, learning will become fun using the puzzle.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the research
* Being 18 years of age or older
* Being a first year student
* Taking the Basic Concepts and Philosophy in Nursing course for the first time
* Not being a student who came via horizontal or vertical transfer
* Not having taken Roper Logan and Tierney's Life Model for Life Activities course
* Not having been absent on the dates when the research data will be collected

Exclusion Criteria:

* Not volunteering to participate in the research
* Being under 18 years old
* Not being a first year student
* Being a student who came via horizontal or vertical transfer
* Being a health vocational high school graduate
* Being a student in the intervention group who did not solve the puzzles
* Being a student in the control group who reached the puzzle booklet and were found to have solved the puzzles.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Personal Information Form | 10 minutes
  This form was prepared by the researchers in line with the literature and includes questions questioning the demographic characteristics of the students such as age, gender, socioeconomic level, etc. This form was used before the training.
Achievement Test 1 | 20 minutes
  It consists of 25 multiple choice questions on the topic of "Roper, Logan, and Tierney's Life Model for Life Activities". This form was used before the training.
Motivation Scale for Instructional Material | 10 minutes
  It was used to measure motivations regarding instructional material. The scale was a 33-item, 5-point Likert type. The highest score that was obtained from the entire scale was 165, and the lowest score was 33. This form was used before and after the training.
Achievement Test 2 | 20 minutes
  It consists of 25 multiple choice questions on the topic of "Roper, Logan, and Tierney's Life Model for Life Activities". This form was used after the training.

CONTACTS AND LOCATIONS:
Locations (1):
- Tarsus University, Mersin, Tarsus, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No